CLINICAL TRIAL: NCT04218981
Title: Definitive Selection of Neuroimaging Biomarkers for the Diagnosis and Treatment to Common Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Guo Wenbin, professor, Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 81771447
Record Dates: First submitted 2019-12-27; First posted 2020-01-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Common Mental Disorder
Keywords: schizophrenia; bipolar disorder; neuroimaging; major depressive disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major | interventions — Antipsychotic Agents; Magnetic Resonance Spectroscopy; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Schizophrenia group (Experimental): 1. Schizophrenia was diagnosed using the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
  2. MRI scan and evaluation of clinical symptoms at baseline and 8 weeks
  3. Choose one of the antipsychotics drugs treatment( olanzapine, risperidone, aminosulpiride) according to the patient's condition
  Interventions: Drug: Antipsychotic drugs
- Bipolar disorder group (Experimental): 1. Bipolar disorder was diagnosed using the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
  2. MRI scan and evaluation of clinical symptoms at baseline and 8 weeks
  3. Choose one of the mood stabilizer drugs treatment( lithium, valproate) according to the patient's condition
  Interventions: Drug: Mood stabilizer
- Major depressive disorder group (Experimental): 1. Major depressive disorder was diagnosed using the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
  2. MRI scan and evaluation of clinical symptoms at baseline and 8 weeks
  3. Choose paroxetine treatment
  Interventions: Drug: Paroxetine
- Healthy controls (No Intervention): MRI scan at baseline and no drugs treatment

INTERVENTIONS:
Drug: Antipsychotic drugs — Choose one of these antipsychotics (olanzapine, risperidone; amisulpride) for schizophrenia group
  Other Names: MRI scan
  Arms: Schizophrenia group
Drug: Mood stabilizer — Choose lithium or valproate for bipolar disorder group
  Other Names: MRI scan
  Arms: Bipolar disorder group
Drug: Paroxetine — Patients with major depressive disorder are treated with paroxetine
  Other Names: MRI scan
  Arms: Major depressive disorder group

SUMMARY:
To explore the whole-brain anatomical and functional abnormalities in drug-naive patients with schizophrenia ,drug-naive patients with BD, drug-naive patients with MDD and healthy controls by using a combination of cross-sectional and longitudinal study designs, including a longitudinal study with 8 weeks of drugs treatment. And explore whether there are shared imaging biomarkers between these three common mental disorders.

DETAILED DESCRIPTION:
Previous studies suggest that there are brain anatomical and functional abnormalities in patients with schizophrenia, bipolar disorder(BD), major depressive disorder(MDD), and the pathogenesis of these three mental disorders may exist overlaps. However, it remains unclear whether these abnormalities can be used for the diagnosis and prediction of treatment effects in mental disorders. It is also unclear whether there are shared imaging biomarkers between these three common mental disorders. In a word, there still lacks reliable neuroimaging biomarkers in mental disorders. Based on the previous studies, this study aims to examine the whole-brain anatomical and functional abnormalities in drug-naive patients with schizophrenia ,drug-naive patients with BD, drug-naive patients with MDD and healthy controls by using a combination of cross-sectional and longitudinal study designs, including a longitudinal study with 8 weeks of drugs treatment( schizophrenia patients are treated with one antipsychotic drug(olanzapine, risperidone; amisulpride); patients with bipolar disorder are treated with one mood stabilizer(lithium;valproate);patients with major depressive disorder are treated with paroxetine). First, neuroimaging biomarkers are definitively selected in patients with different mental disorders for the purpose of diagnosis by using a cross-sectional design. After that, a longitudinal study is conducted in patients after 8 weeks of drugs treatment to validate that the selected neuroimaging biomarkers can be used to predict treatment response of medication. The definitively selected neuroimaging biomarkers are expected to be useful for the diagnosis and prediction of treatment effects in these three mental disorders; and therefore to be helpful for understanding the pathophysiology of mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for schizophrenia,bipolar disorder, major depressive disorder according to the Structural Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Never received any treatment before.
* For healthy controls: their first-degree relative had no history of psychiatric disorders.

Exclusion Criteria:

* The exclusion criteria for all subjects were as follows: any physical illnesses, such as liver, kidney, and cardiovascular diseases; any current or past neuropsychiatric disorders; any traumatic brain injury; seizures; serious impulsive behavior; drug or alcohol addiction; contraindications for MRI; and pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Resting-state functional magnetic resonance imaging (fMRI) data acquisition for all participants | 8 week
  A 3.0 T Siemens scanner (Germany) was applied to obtain the MRI images in the Second Xiangya Hospital of Central South University.The MRI data will be obtained before and after treatment at different follow up point.All participants were told to lie on the scanner with their eyes closed. They wore soundproof headphones and asked to remain still. The parameters were as follows: repetition time of 2710 ms, echo time of 3.78 ms, flip angle of 7°, inversion time of 1000 ms, slice thickness of 1 mm, field of view of 256 mm × 256 mm, matrix of 256 × 256, no gap, and 188 slices.
Positive and Negative Syndrome Scale (PANSS) | 8 week
  The PANSS total scores ,subscale scores were used to evaluate the severity of psychotic symptoms at baseline and eight weeks for schizophrenia.The total score of the PANSS was more than 60.The higher scores mean a worse outcome.
Hamilton Depression Scale-17 (HAMD-17) | 8 week
  HAMD-17 total scores were used to evaluate the severity of depressive symptoms at baseline and eight weeks for major depressive disorder. The total score of the HAMD-17 was more than 17.The higher scores mean a worse outcome.
Young Mania Rating Scale (YMRS) | 8 week
  YMRS total scores were used to evaluate the severity of manic symptoms for bipolar disorder before and after treatment at different follow up point.The higher scores mean a worse outcome.
Brief Cognitive Assessment Tool for schizophrenia(B-CATS) | 8 week
  The investigators will use the B-CATS scale to assess cognitive function before and after treatment at different follow up point.The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Social Disability Screening Schedule(SDSS) | 8 week
  The investigators will use the SDSS scale to assess social function before and after treatment at different follow up point.The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Guo, Study Director — The Second Xiangya Hospital, Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China